CLINICAL TRIAL: NCT04557826
Title: A Phase I Open-label, First-in-Man Acute Safety, Tolerability and Device Acceptability Study of Experimental Device RD19 for Protection From Human Respiratory Tract Pathogens
Brief Title: Acute Safety and Acceptability Study of Experimental Device RD19 for Protection From Human Respiratory Disease Pathogens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EmitBio Inc. (Industry)
Responsible Party: Sponsor
Organization: KNOWBio Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RD19-01-Q320
Record Dates: First submitted 2020-08-31; First posted 2020-09-22 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- RD19 Experimental Device (Experimental): RD19 Experimental Device used twice/day for 3 minutes each use at least 4 hours, and preferably 8-12 hours, apart
  Interventions: Device: RD19

INTERVENTIONS:
Device: RD19 — Experimental device that uses safe electromagnetic energy to stimulate the proximal repository of respiratory tract infectious disease pathogens

SUMMARY:
This first-in-man (FIM) phase I study will evaluate the acute safety, tolerability, and acceptability of the investigational RD19 device among 25 healthy volunteers between the age of 18 and 45.

DETAILED DESCRIPTION:
This first-in-man (FIM) phase I study will evaluate the acute safety, tolerability,and acceptability of the investigational RD19 device among 25 healthy volunteers between the age of 18 and 45. Based on the results of numerous preclinical studies, a short 3 minute use twice a day, separated by at least 4 hours, preferably 8 to 12 hours apart) will be evaluated.

Safety and tolerability (local reactogenicity) will be assessed actively at the following study days: screening (baseline set), 1, 7 and 14, and on non-clinic visit days by collection of these data by history during clinic visits via a memory aid (diary cards). Volunteers will be encouraged to promptly contact designated clinical trial staff or the one of the Sponsor's Emergency Response Team for AEs of a medically urgent nature.

A Comprehensive Metabolic Panel, as well as CBC with differential, urinalysis, and pregnancy testing will be performed at screening and at Day 14 or early termination (and potentially during unscheduled) clinic visits. Hematological safety assessments (evaluation of methemoglobinemia) will be performed at all visits.

Study volunteers will be asked to immediately contact the clinical coordinator and/or the PI in all instances where they experience an AE of greater than moderate intensity. Volunteers will be instructed to report to the clinical trial unit for an unscheduled visit or to seek the appropriate level of medical care based on the nature of their AE/SAE. In all such instances, all relevant information pertaining to these significant medical events will be captured on the appropriate e-CRFs.

Hematology safety laboratory evaluations will be performed at screening, as well during all scheduled clinic visits. Laboratory assessments may be part of the evaluation of medically attended AE evaluation and for all SAEs.

Upon ratification of the CTA, the site began pre-recruitment outreach efforts of potential volunteers within M3-WRA's database to ascertain "interest in general" in this study. Official recruitment which may include fliers, letters, telephone calls, etc. and specific recruitment of potential subjects who have previously participated in other clinical studies conducted at the site commenced only after formal IRB approval. Other forms and/or mechanisms of recruitment may also be used. The IRB will approved the recruitment process and all materials prior to use.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to initiation of any study
2. Agrees to comply with planned study procedures and be available for all study visits.
3. Agrees to the collection of venous blood per protocol.
4. Male or non-pregnant female, 18 to 45 years of age, inclusive, at time of enrollment.
5. Body Mass Index 18-35 kg/m2, inclusive, at screening.
6. Woman of childbearing potential must have a negative urine pregnancy test within 7 days prior to study initiation.
7. Oral temperature is less than 100.0°F (37.8°C).
8. Pulse no greater than 90 beats per minute.
9. Systolic BP is 85 to 150 mmHg and Diastolic BP ≤ 90 mmHg, inclusive.
10. Clinical screening laboratory evaluations are within acceptable normal reference ranges at the clinical laboratory being used.

Exclusion Criteria:

1. Positive urine pregnancy test at screening.
2. Has any medical disease or condition that, in the opinion of the site PI or appropriate sub- investigator, precludes study participation.
3. Plans to travel away from the study site area during the term of study to a location or in a manner that may interfere with full completion of the study per protocol.
4. Presence of self-reported or medically documented significant medical or psychiatric condition(s).
5. Has an acute illness, as determined by the site PI or appropriate sub-investigator, with or without fever [oral temperature >37.8°C (100.0°F)] within 72 hours of study day 1.
6. Reports a recent positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or HIV-1 antibodies at screening.
7. Currently enrolled in or plans to participate in another clinical trial with an interventional investigational agent that will be received during the study period.
8. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to nitrates, nitrites or sun exposure.
9. Active use of any medications that may be associated with pharyngeal or oral mucosal irritation.
10. Has any blood dyscrasias or significant disorder of coagulation.
11. Has a history of alcohol abuse or other recreational drug (excluding cannabis) use within 1 month of Study Day 1.
12. Has any oral abnormality that would interfere with device use, or intra-oral metal body piercings that cannot be removed for the duration of the study. Metal orthodontia is permitted as braces will be covered by the device mouthpiece.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Cohen, DO, Principal Investigator — M3-Wake Research Associates Carolina Phase I
Locations (1):
- Carolina Phase I, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RD19 Experimental Device
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RD19 Experimental Device
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: RD19 Acceptability
Description: * Ease of device use (Likert Scale 1 -10)
  * Clarity of user instructions (Likert Scale 1-10)
  * Compliance with per protocol schedule (# times missed / 28) and, if out of compliance, reason(s) for noncompliance (collected as verbal string).
Time Frame: 14 consecutive days of RD19 device use per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | RD19 Experimental Device
Number analyzed (Participants) | 25
Participants
  I Did Not Have Any Problems Using The Device Full Assessment Period (Day 7): Strongly Disagree | 1
  I Did Not Have Any Problems Using The Device Full Assessment Period (Day 7): Disagree | 0
  I Did Not Have Any Problems Using The Device Full Assessment Period (Day 7): Neutral | 1
  I Did Not Have Any Problems Using The Device Full Assessment Period (Day 7): Agree | 9
  I Did Not Have Any Problems Using The Device Full Assessment Period (Day 7): Strongly Agree | 13
  I Did Not Have Any Problems Using The Device Full Assessment Period (Day 7): Not recorded | 1
  I Did Not Have Any Problems Using The Device Full Assessment (Day 14): Strongly Disagree | 0
  I Did Not Have Any Problems Using The Device Full Assessment (Day 14): Disagree | 2
  I Did Not Have Any Problems Using The Device Full Assessment (Day 14): Neutral | 0
  I Did Not Have Any Problems Using The Device Full Assessment (Day 14): Agree | 6
  I Did Not Have Any Problems Using The Device Full Assessment (Day 14): Strongly Agree | 15
  I Did Not Have Any Problems Using The Device Full Assessment (Day 14): Not recorded | 2

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | RD19 Experimental Device
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 14/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RD19 Experimental Device (N=25)
Headache (Nervous system disorders) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Oral Disorder (Gastrointestinal disorders) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dry throat (Gastrointestinal disorders) | 1 (1)
Application Site Pain (General disorders) | 6 (6)
Application Site Erythema (General disorders) | 4 (4)
Application Site Swelling (General disorders) | 1 (1)
Dizziness (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a phase I, open-label, safety study and is not designed to test any statistical hypotheses. Rather, this is a descriptive study intended to obtain preliminary estimates in healthy adults of the safety, including reactogenicity, of the EmitBio™ RD19 Device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data and reports of study data are the property of the study sponsor. The sponsor my grant the PI the right to publish the results of this research in a scientific journal, conditional upon the review and concurrence of the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT04557826/Prot_SAP_000.pdf